CLINICAL TRIAL: NCT06322316
Title: Analgesic Efficacy of Ultrasound-guided Retrolaminar Block and Erector Spinae Plane Block in Modified Radical Mastectomy: A Randomized Controlled Study
Brief Title: Analgesic Efficacy of U/S Retrolaminar Block and Erector Spinae Plane Block in MRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Soliman, lecturer of anesthesia, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-492-2022
Record Dates: First submitted 2024-03-05; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms; Analgesia
Keywords: Analgesics; Opioids; Breast Neoplasms; Postoperative Pain; Mastectomy; Nerve block
MeSH Terms: conditions — Breast Neoplasms; Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: To determine the analgesic effect of ultrasound guided Retrolaminar Block and Erector Spinae Plane Block in patients undergoing modified radical mastectomy regarding the following : 1-Post-operative opioid (morphine) consumption in the 1st 24 hours 2- Postoperative Numeric Pain Rating Scale. 3. Effect on hemodynamics: Mean arterial blood pressure and Heart rate. 4. Intraoperative fentanyl consumption. 5. Duration of analgesic effect
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 30 patients. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Ultrasound-guided Retrolaminar Block (RLB) Group (Active Comparator): Received a preoperative ultrasound-guided retrolaminar block using 20 ml levobupivacaine 0.25% Ultrasound probe was placed on the back in a transverse orientation on the lateral side of the posterior median line to identify the lamina of the 5th vertebra, ESM, and transversospinalis muscles of the target segment.
  Interventions: Procedure: The Ultrasound-guided Retrolaminar Block Group
- The Ultrasound-guided Erector Spinae Plane Block (ESPB) Group (Active Comparator): Received a preoperative ultrasound-guided erector spinae plane block using 20 ml levobupivacaine 0.25%.
  ultrasound probe was placed on the back in a transverse orientation to identify the tip of the T5 transverse process as flat, squared-off acoustic shadows with a faint image of the pleura visible. When the tip of the transverse process was centered on the ultrasound screen, the probe was rotated to a longitudinal orientation. In the parasagittal view The block needle was inserted in-plane in a cranial-to-caudal direction until contact was made with the T5 transverse process.
  Interventions: Procedure: The Ultrasound-guided Erector Spinae Plane Block Group

INTERVENTIONS:
Procedure: The Ultrasound-guided Retrolaminar Block Group — The ultrasound probe was placed on the back in a transverse orientation on the lateral side of the posterior median line to identify the lamina of the 5th vertebra, ESM, and transversospinalis muscles of the target segment.
  A 38-mm 22-gauge regional block needle was advanced using an in-plane technique. When the puncture needle touched the lamina, 20 mL of 0.25% levobupivacaine was administered between the transversospinalis muscle and lamina. The LA diffusion between the lamina and the ESM indicated a successful puncture.
  Other Names: RLB
  Arms: The Ultrasound-guided Retrolaminar Block (RLB) Group
Procedure: The Ultrasound-guided Erector Spinae Plane Block Group — The ultrasound probe was placed on the back in a transverse orientation to identify the tip of the T5 transverse process as flat, squared-off acoustic shadows with a faint image of the pleura visible. When the tip of the transverse process was centered on the ultrasound screen, the probe was rotated to a longitudinal orientation. In the parasagittal view, the following layers were visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius, ESM, and T5 transverse process.
  The block needle was inserted in-plane in a cranial-to-caudal direction until contact was made with the T5 transverse process. The correct location of the needle tip in the fascial plane deep to the ESM was confirmed by injecting 0.5-1.0 ml of normal saline and seeing the fluid lifting the ESM off the transverse process without distending the muscle. Then 20 ml levobupivacaine 0.25% was injected.
  Other Names: ESPB
  Arms: The Ultrasound-guided Erector Spinae Plane Block (ESPB) Group

SUMMARY:
Modified radical mastectomy (MRM) is the most commonly performed surgical procedure in breast cancer patients and is usually associated with severe postoperative pain. The peripheral nerve block techniques were suggested to reduce acuter post-mastectomy pain. The study compared the analgesic efficacy of retrolaminar block (RLB) and ESPB in patients undergoing MRM.

DETAILED DESCRIPTION:
Introduction Globally, breast cancer remains the most prevalent cancer among females, with an estimated incidence of 31% and mortality of 15%. Surgery is foremost in managing breast cancer, where modified radical mastectomy (MRM) is the most commonly performed procedure. This procedure implicates vigorous tissue dissection and seroma formation with many postoperative complications. Pain is the main complaint following MRM, affecting up to 50% of women, and 25-60% develop persistent chronic postmastectomy pain.

Therefore, adequate pain control is crucial to postoperative management after MRM. Numerous analgesic methods were suggested to reduce acuter post-mastectomy pain. Opioid-related adverse events include nausea and vomiting, respiratory depression, sedation, and dizziness.

Most mastectomy-related pain originates from the chest wall's sensory nerves. The peripheral nerve block techniques have gained increased interest in treating postoperative pain. The erector spinae plane block (ESPB) is one of these techniques that proved effective in various surgical procedures, including breast surgery. It encompasses injecting the local anesthetic (LA) solution deep into the erector spinae muscle (ESM), which eventually spreads through the paravertebral space. Ultrasound-guided retrolaminar block (RLB) is another approach that was found to be effective for pain relief after thoracic surgery. In RLB, LA is injected into the space between the ESM and the lamina of the thoracic vertebra.

Both techniques are considered variants of paravertebral block; however, prospective studies comparing RLB and ESPB are limited. Therefore, this study was designed to compare the analgesic efficacy of ultrasound-guided retrolaminar block and erector spinae plane block in patients undergoing modified radical mastectomy.

Patients and Methods:

This randomized single-blinded study was conducted at the National Cancer Institute (NCI), Cairo University from October 2022 and finished March 2023. The study was approved by the institutional review board and the scientific committee of the anesthesia department of the NCI and Faculty of Medicine, Cairo University. All participants provided written informed consent before enrollment in the study after fully explaining the procedures and possible complications.

The study involved 60 female patients scheduled for MRM under general anesthesia with the following inclusion criteria: age 18 to 65, ASA class II or III, and body mass index (BMI) of 20-35 kg/m2. Patients with known sensitivity or contraindication to the drugs used in the study, history of psychological disorders or chronic pain syndromes, contraindication to regional anesthesia (local sepsis, pre-existing peripheral neuropathies, coagulopathy), severe respiratory or cardiac conditions, advanced liver or kidney disease were excluded from the study.

The patients were randomly allocated into one of two equal groups using computer-generated random numbers in opaque closed envelopes. An independent statistician performed the randomization. The grouping was revealed only when the patient was transferred to the pre-anesthetic room. The RLB Group (n=30) received a preoperative ultrasound-guided retrolaminar block using 20 ml levobupivacaine 0.25%. The ESPB Group (n=30) received a preoperative ultrasound-guided erector spinae plane block using 20 ml levobupivacaine 0.25%.

Preoperative assessment included thorough history taking, physical examination, and laboratory and radiological investigations. The patients were instructed to report pain using the Numeric Pain Rating Scale (NPRS), where 0 = no pain and 10 = worst imaginable pain. All patients were premedicated with IV midazolam 0.01-0.02 mg/kg 30 minutes before surgery. In both blocks, a Fujifilm Sonosite M-Turbo Ultrasound system linear probe was used (SN.04RQZ6) . After performing blocks lung ultrasound was performed to exclude pneumothorax.

Retrolaminar Block Technique The block was performed under complete aseptic precautions. The ultrasound probe was placed on the back in a transverse orientation on the lateral side of the posterior median line to identify the lamina of the 5th vertebra, ESM, and transversospinalis muscles of the target segment. A skin wheal using 3 ml of 1% lidocaine was made 2-3 cm medial to the transducer. A 38-mm 22-gauge regional block needle was advanced using an in-plane technique. When the puncture needle touched the lamina, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% levobupivacaine was administered between the transversospinalis muscle and lamina. The LA diffusion between the lamina and the ESM indicated a successful puncture.

Erector spinae plane block:

The ultrasound probe was placed on the back in a transverse orientation to identify the tip of the T5 transverse process as flat, squared-off acoustic shadows with a faint image of the pleura visible. When the tip of the transverse process was centered on the ultrasound screen, the probe was rotated to a longitudinal orientation. In the parasagittal view, the following layers were visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius, ESM, and T5 transverse process. A skin wheal was made using 3 ml of 1% lidocaine; then, the block needle was inserted in-plane in a cranial-to-caudal direction until contact was made with the T5 transverse process. The correct location of the needle tip in the fascial plane deep to the ESM was confirmed by injecting 0.5-1.0 ml of normal saline and seeing the fluid lifting the ESM off the transverse process without distending the muscle. After aspiration to avoid intravascular injection, 20 ml levobupivacaine 0.25% was injected.

Anesthetic Management:

All patients were monitored continuously using electrocardiography, non-invasive blood pressure, peripheral O2 saturation, temperature probe, and end-tidal CO2 throughout the surgical procedure. Anesthesia was induced using fentanyl 2 μg/kg and propofol 2 mg/kg IV. Tracheal intubation was facilitated using rocuronium 0.5 mg/kg IV. Anesthesia was maintained with inhaled sevoflurane 2.0-2.5% in oxygen-enriched air (FiO2=0.5). Maintenance doses of rocuronium 0.1 mg\kg were provided every 30 minutes. Paracetamol 500 mg and ketorolac 30 mg were provided as a part of multimodal analgesia. Rescue analgesia of fentanyl 1 μg/kg was given if the mean arterial blood pressure (MAP) or heart rate (HR) rose above 20% of baseline levels. The patients were mechanically ventilated at appropriate settings to keep end-tidal CO2 at 30-35 mmHg.

The first reading of MAP and HR was taken before induction of general anesthesia as a baseline reading. Then, another reading was taken immediately before incision and at 30-minute intervals intraoperatively. Hypotension (reduction > 20% of baseline reading) was treated with 0.9% normal saline and/or 5 mg ephedrine in incremental doses to maintain MAP above 70 mmHg. The residual neuromuscular blockade was reversed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Extubation was performed after complete recovery of the airway reflexes.

Postoperatively the NPRS score, MAP, and HR were noted immediately on arrival and every 2 hours. Multimodal analgesia was provided as paracetamol 500 mg/6 hours and ketorolac 30 mg/8 hours IV. Rescue analgesia was provided as IV morphine 3 mg boluses when the patient indicated an NPRS score ≥ 4. The total amount of morphine given in 24 hours was recorded, and a maximum dose of 0.5 mg/kg/24 hours of morphine was allowed. Side effects such as nausea, vomiting, sedation, hallucination, and respiratory depression (respiratory rate < 10/minute) were recorded. Moderate or severe postoperative nausea and vomiting (PONV) was treated with 0.1 mg/kg of IV ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Type of surgery; Modified Radical Mastectomy (MRM)
* Physical status ASA I, II, III.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Age <18 years or >65 years
* BMI <20 kg/m2 and >35 kg/m2
* Known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.
* Pregnancy.
* Physical status ASA IV and Male patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
the total morphine consumed postoperatively for 24 hours | 24 hours
  the total morphine consumed postoperatively for 24 hours

SECONDARY OUTCOMES:
the total intraoperative fentanyl consumption | intraoperative
  the total intraoperative fentanyl consumption when hemodynamics intraoperative >20%
duration of analgesia | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Duration of analgesia was defined as the time from the block performance to the first postoperative rescue analgesic administrated upon patient request
postoperative nausea and vomiting PONV as side effect of morphine | at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively
  nausea and vomiting scores using a four-point verbal scale

CONTACTS AND LOCATIONS:
Locations (1):
- National cancer Insititute Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
till publication